CLINICAL TRIAL: NCT00795587
Title: Compared Effects of 2 Doses of Mannitol on Post Traumatic Intracranial Hypertension
Brief Title: Comparison of 2 Doses of Mannitol on Post Traumatic Intracranial Hypertension and Cerebral Monitoring
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: evolution of patient's care allows no more recruitment
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0816; 2008-004979-21 (EudraCT Number)
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-11

CONDITIONS: Traumatic Brain Injury; Intracranial Hypertension
MeSH Terms: conditions — Brain Injuries, Traumatic; Intracranial Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mannitol high dose (Active Comparator): mannitol 20% 0,8 g/ kg on minutes
  Interventions: Drug: variation of mannitol dose
- mannitol low dose (Active Comparator): mannitol 20% 0,4 g/ kg on minutes
  Interventions: Drug: variation of mannitol dose

INTERVENTIONS:
Drug: variation of mannitol dose — in case of intracranial hypertension up to 20 mmHg lasting more than 10 minutes and without nociceptive stimulation or systemic instability: injection of either 0.4 g/ kg or 0.8 g/ kg of mannitol 20% (randomized) on 20 minutes, with monitoring of neurologic, systemic and biologic datas during 120 minutes

SUMMARY:
Will an increase of the dose of mannitol improve the effects on neuromonitoring in patients suffering intracranial hypertension following traumatic brain injury?

DETAILED DESCRIPTION:
traumatic brain injury intracranial hypertension 0,4 g/ kg vs 0,8 g/ kg (randomized) on 20 minutes monitoring: ICP, transcranial doppler, brain pO2, MAP, HR, diuresis, biology duration: 2 hours

ELIGIBILITY:
Inclusion Criteria:

* adults
* severe traumatic brain injury
* intracranial hypertension requiring mannitol administration

Exclusion Criteria:

* impeding neurosurgery
* hemodynamic or respiratory severe failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
intracranial pressure | 2 hours

SECONDARY OUTCOMES:
transcranial doppler | 2 h
brain PO2 | 2h
MAP | 2h
Heart Rate | 2h
biology (blood gases, natremia, hematocrit) | 2h
diuresis | 2h
fluid requirement | 2h

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Francony, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Universitary Hospital, Grenoble, France